CLINICAL TRIAL: NCT05282134
Title: Comparison of the Effectiveness of Wet Cupping and Acupuncture in Migraine: A Randomized Controlled Study
Brief Title: Comparison of Wet Cupping and Acupuncture in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Head of the complementary medicine department, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCTACCU1
Record Dates: First submitted 2022-03-05; First posted 2022-03-16 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Migraine
Keywords: Migrain, Wet Cupping, Acupuncture, VAS, MIDAS
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wet cupping therapy (Experimental): The intervention group will undergo 3 successive wet cupping therapy (WCT) sessions once in a month throughout 3 months (On 0, 30, and 60 days. Cups will be held for 5 minutes on the 5 regions of the C7 cervical spine (DU14 acupuncture point), bilateral T2-4 lateral spine (BL41-42 acupoint) and bilateral T6-8 lateral spine (BL44-46) points, which are recommended areas for headache, Then, these areas where the blood supply has increased will be drawn with a sterile lancet and the cup will be applied again and left for 10 minutes, and then the cups will be removed and the accumulated blood will be cleaned.
  Interventions: Procedure: Wet cupping therapy
- Acupuncture (Experimental): Acupuncture application will be done by manually needling selected acupuncture points specific to the disease twice a week for 4 weeks. After the needles are placed, they will be manipulated to create a feeling of de-qi and left for 20 minutes.
  Interventions: Procedure: Acupuncture
- Control (No Intervention): Control group will not receive any intervention

INTERVENTIONS:
Procedure: Wet cupping therapy — Wet cupping therapy is a bloodletting application done by cups on the skin
  Other Names: Hijama
  Arms: Wet cupping therapy
Procedure: Acupuncture — Acupuncture is a complementary application of TCM done by needles
  Arms: Acupuncture

SUMMARY:
The aim of this study is to evaluate the effects of wet cupping therapy (WCT) on migraine patients and compare it with acupuncture. The patients will be randomized into three groups. WCT will be applied once a month to patients in group 1 and acupuncture will be applied to group 2, while the control group (group 3) will be on standard therapy for migraine. An evaluation will be made before treatment and at the 3rd month using the MIDAS and VAS.

DETAILED DESCRIPTION:
Background: The most common primary headache is migraine. Migraine was ranked as the sixth cause of years lost due to disability all over the world in 2013. . About 15% of the world's population has migraine. Every year, 14-35% of women and 6-15% of men have migraine. The economic burden caused by the disease, which is so common and affects new masses every year, is substantial, as well as the loss of workforce, treatment costs. According to the UK-NHS data; Migraines cause an economic burden of 2.25 billion pounds based on 25 million lost days each year and more than 150 million pounds based on care, examinations, and treatment. There may be some side effects, drug interactions, comorbid conditions, and resistance cases in pharmacological treatments. In this context, traditional treatment methods may be preferred due to the low incidence of side effects. . In this context, traditional treatment methods may be preferred due to the low incidence of side effects. Acupuncture, which is widely used among traditional methods, has been shown to reduce the frequency of headaches. There are few studies on the effectiveness of Hijama, which is another traditional method and frequently used in our geography,

Purpose: The aim of the study is to investigate and compare the efficacy of wet cupping and acupuncture therapies in patients with migraine

Method: The patients who were referred to Umraniye Training Hospital Neurology polyclinic and diagnosed with migraine will be enrolled in the study.

The inclusion criteria are being 18-65 years old, having been diagnosed with migraine (ICHD-3 diagnosis criteria), and consenting to participate in the study. Those who are accompanied with any chronic disease and on daily medication, contraindicated to WCT as determined in the routine blood tests that were routinely performed before the prior to application (Hgb <9,5; INR> 1,2,; Hgb <9,5, etc) and who received WCT in the last three months will be excluded.

The volunteers will be randomized into three separate groups as wet cupping, acupuncture, and control group Control group will not receive any intervention. The wet cupping group will undergo 3 successive WCT sessions once in a month throughout 3 months (On 0, 30, and 60 days). Vacuum cups will be used on different acupuncture points to perform WCT: The one on the posterior median line, in the depression below the processus spinosus of the 7th cervical vertebra, was DU 14 (Dazhui) point; the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 3rd thoracic vertebra interscapulum region were UB 42 (Pohu) bilateral points; and the ones on the back, 3.0 cm lateral to the lower border of the spinous process of the 7th thoracic vertebra were UB 46 (Geguan) bilateral points and additionally the patient's trigger points which we detect during the examination. There will be 5-7 points in total. The technique used will be triple S (Sucking, Scarification, Sucking) in all sessions.

The acupuncture group will receive acupuncture application which will be done by manually needling on selected acupuncture points specific to the disease twice a week for 4 weeks. After the needles are placed, they will be manipulated to create a feeling of de-qi and will be left for 20 minutes.

At 0 and 3 months, MIDAS and VAS questionnaires will be applied to all patient groups Evaluation and comparison between the groups will be made with the scores of these questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65 who were diagnosed with migraine, no concomitant chronic disease and who gave their consent to participate in the study will be recruited.

Exclusion Criteria:

* 1. Having a bleeding diathesis

  2. Receiving antithrombotic and antiaggregant therapy

  3. Chronic disease that requires continuous drug use have

  4. Wet cupping or hirudotherapy treatment in the last 3 months to have received 5.Be younger than 18 years old and over 65 years old 6. Having a hemoglobin value below 9.5 g/dl 7. INR value over 1.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The change from the baseline (at 0 month) MIDAS scores at 3th month | At 0 and 3 months
  The Migraine Disability Assessment (MIDAS) questionnaire is a brief, self-administered questionnaire designed to quantify headache-related disability over a 3 month period.
The change from the baseline (at 0 month) VAS scores at 3 th month | At 0 and 3 months
  Visual analogue scales (VAS) are well-validated instruments for assessing pain intensity. Scores are recorded by a mark on a 10-cm line that represents 0 as "no pain" and 10 as "worst pain."

CONTACTS AND LOCATIONS:
Overall Officials: Emin Pala, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, İ̇stanbul, Turkey (Türkiye)